CLINICAL TRIAL: NCT05602558
Title: A Randomized, Double-blinded, Placebo-controlled Phase II/III Clinical Trial to Evaluate the Efficacy, Safety and Immunogenicity of a Recombinant SARS-CoV-2 Vaccine (CHO Cell) LYB001 as Booster Vaccination in Adults 18 Years of Age or Older Completed Two-dose or Three-dose Inactivated COVID-19 Vaccine
Brief Title: The Phase Ⅱ/Ⅲ Trial of LYB001
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yantai Patronus Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LYB001/CT-PAK-301
Record Dates: First submitted 2022-10-21; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LYB001 (Experimental)
  Interventions: Biological: LYB001
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: LYB001 — The antigen consists of receptor-binding domain (RBD) from wild-type SARS-CoV-2 displaying on virus-like particle (VLP) vector, adjuvanted with aluminium hydroxide.
  Arms: LYB001
Biological: Placebo — Aluminium hydroxide adjuvant
  Arms: Placebo

SUMMARY:
The study will be conducted in two phases using a randomized, double-blind, placebo-controlled design. A phase II trial will be initiated to assess the safety of LYB001 as booster shots, and then proceed to a phase III trial to assess the vaccine efficacy (VE) of LYB001 against COVID-19 after an acceptable safety profile, per the judgement of Data and Safety Monitoring Board (DSMB), within 28 days after booster in the phase Ⅱ trial is assessed. After collection of 155 COVID-19 cases, all participants will get unblinded. Participants assigned to the placebo group can choose to receive LYB001 vaccine at their own discretion.

Phase II stage:

The purpose of phase Ⅱ study is to assess the safety of healthy subjects aged 18 years and older who have completed two-dose or three-dose inactivated COVID-19 vaccine for 6-18 months. About 200 age s-stratified subjects aged over 18 years will be randomly assigned to receive the LYB001 or placebo in a 1:1 ratio in the deltoid muscle of the upper arm.

The Phase III study will be initiated after the DSMB confirm that all subjects in Phase II experience acceptable safety profile within 28 days after booster. All subjects in Phase II trial will be required to complete efficacy follow-ups for 12 months along with safety observation, and will be included in the Phase III efficacy analysis set (Phase II data will eventually be combined with Phase III data for statistical analysis, including efficacy and safety data).

Phase III stage:

A total of 17800 participants aged 18 years and older who have completed two-dose or three-dose inactivated COVID-19 vaccine for 6-18 months. The participants will be randomly assigned to the LYB001 booster or placebo booster group in 1:1 ratio according stratification factors of study center and age (18-59 years vs. ≥60 years) , with participants aged ≥ 60 years accounting for over 20 percent of total population.

After booster vaccination, all subjects will be evaluated for protective efficacy and safety, and 1000 subjects (800 subjects aged 18-59 years, and 200 subjects aged ≥60 years) will be enrolled in the subgroup for immunogenicity evaluation (LYB001: Placebo=1:1).

All subjects will be followed up to 12 months after booster vaccination. The entire clinical study will be completed after the pre-defined COVID-19 cases has been achieved and each participant has completed 12-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 18 years and older, including both males and females;
* Subjects who agree to participate in this clinical trial voluntarily and sign the informed consent form, are capable of providing valid identification, understanding and complying with the requirements of the clinical protocol.
* Subjects who have been vaccinated with two-dose or three-dose inactivated COVID-19 vaccine for6-18 months (including boundary values).
* For female participants of childbearing potential, effective contraception measures should be used within 2 weeks prior to participation in this study and the results of pregnancy test is required to be negative. Participants should voluntarily agree to use effective contraceptive measures from the time of signing the informed consent form to the end of the study (effective contraceptive measures including oral contraceptives (excluding emergency contraceptives), injectable or implantable contraceptives, sustained-release topical contraceptives, hormonal patches, intrauterine device, sterilization, abstinence, condoms (for males), diaphragms, cervical caps, etc.).

Exclusion Criteria:

* Receipt of any COVID-19 prophylactic medication other than inactivated COVID-19 vaccine (e.g., receipt history of any approved or under developing COVID-19 vaccines, or other COVID-19 prophylactic medication, etc.), or previous vaccination history other than other than two- or three-dose inactivated COVID-19 vaccination;
* Systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg (for subjects with poorly controlled blood pressure), or axillary body temperature ≥ 37.3°C prior to enrolment;
* Known allergy, or history of anaphylaxis or other serious adverse reactions to vaccines or their excipients;
* History of severe acute respiratory syndrome (SARS) or Middle East respiratory syndrome (MERS);
* History of COVID-19, or positive results for SARS-CoV-2 nucleic acid or antigen tests at screening;
* Receipt of any live attenuated vaccine within 28 days prior to vaccination, and other vaccines such as subunit and inactivated vaccine within 14 days prior to vaccination;
* Receipt of blood or blood-related products, including immunoglobulins, monoclonal antibodies, within 3 months prior to vaccination; or any planned use during the study period.
* Subjects with the following diseases:

  1. Any acute diseases or acute attacks of chronic diseases within 7 days prior to enrolment；
  2. Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.；
  3. Congenital or acquired immunodeficiency or autoimmune disease, or long-term receipt (>14 consecutive days) of glucocorticoid (reference value for dose: ≥20 mg/day prednisone or equivalent) or other immunosuppressive agents within the past 6 months, with exception of inhaled or topical steroids, or short-term use (≤14 consecutive days) of oral corticosteroids；
  4. Currently suffering from or diagnosed with infectious diseases, such as hepatitis B, hepatitis C, syphilis, AIDS etc.；
  5. History or family history of neurological disorders (convulsions, epilepsy, encephalopathy, etc.) or psychiatric disorders；
  6. Asplenia, or functional asplenia；
  7. Presence of severe, uncontrollable or hospitalized cardiovascular diseases, endocrine diseases, blood and lymphatic diseases, immune diseases, liver and kidney diseases, respiratory diseases, metabolic and skeletal diseases, or malignant tumors;
  8. Contraindications to IM injections and blood draws, such as coagulation disorders, thrombotic or bleeding disorders, or conditions that needs continuous anticoagulant usage.
* Drug or alcohol abuse (alcohol intake ≥ 14 units per week) which in the investigator's opinion would compromise the participant's safety or compliance with the study procedures;
* Pregnant or lactating females;
* Having participated or participating in COVID-19 related clinical trials, and those participating or planning to participate in other clinical trials during the study period;
* Presence of any underlying disease or condition which, in the opinion of the investigator, may place the subject at unacceptable risk, is unable to meet the requirements of the protocol, or interfere with the assessment of vaccine response.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18000 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
First occurrence of confirmed symptomatic COVID-19 incidence rate per person-years of follow-up | 14 days after the booster

SECONDARY OUTCOMES:
First occurrence of confirmed severe, critical, and fatal COVID-19 incidence per person-years of follow-up | 14 days after the booster
Solicited local/systemic adverse events | 7 days after the booster
Unsolicited adverse events | 28 days after the booster
Geometric mean titers of neutralizing antibodies against wild-type SARS-CoV-2 and circulating variants of concern, S protein-binding antibodies in immunogenicity subgroup | 14days, 28 days after booster, and 3, 6, 12 months after booster
Geometric mean fold rises of neutralizing antibodies against wild-type SARS-CoV-2 and circulating variants of concern, S protein-binding antibodies in immunogenicity subgroup | 14days, 28 days after booster, and 3, 6, 12 months after booster
Seroconversion rates of neutralizing antibodies against wild-type SARS-CoV-2 and circulating variants of concern, S protein-binding antibodies in immunogenicity subgroup | 14days, 28 days after booster, and 3, 6, 12 months after booster

IPD SHARING:
Plan to Share IPD: No